CLINICAL TRIAL: NCT05717556
Title: Factors Affecting Success of First Attempt in Ultrasonography-Guided Internal Jugular Vein Catheterization
Brief Title: Success of Internal Jugular Vein Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Köksal, Medical Doctor, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/12-6
Record Dates: First submitted 2023-01-31; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Ultrasound; Catheterization; Volume Status
Keywords: juguler vein catheterization; ultrasound guidance; pleth variability index

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single attempt catheterization (Active Comparator): successful catheterization with a single attempt number
  Interventions: Procedure: Internal Jugular Vein Catheterization
- multiple attempts catheterization (Active Comparator): successful catheterization after multiple attempts
  Interventions: Procedure: Internal Jugular Vein Catheterization

INTERVENTIONS:
Procedure: Internal Jugular Vein Catheterization — Inserting a cannula into the internal jugular vein

SUMMARY:
Internal jugular vein cannulation can be performed with the blind technique under ultrasound (USG) guidance or using classical marker points. It has been shown that USG-guided interventions reduce the complication rate compared to the method performed with the blind technique (4%/13.5%). In addition, the initial entry success rate in the USG supported group is 65%. , this rate remained at 45% with the blind technique.

Although Pleth variability index monitoring is a noninvasive method, it is a technique that consistently predicts fluid sensitivity in patients under mechanical ventilation.

The aim of study is before applying USG guided catheterization; We think that by revealing the factors of the patient that are effective on the number of interventions, necessary measures can be taken for the success of catheterization as a result.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-75
* underwent coronary artery bypass surgery

Exclusion Criteria:

* <18 years old
* Hemodynamic instability
* Use of inotropic agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
factors of internal vein jugular catheterization success | Baseline (Before catheterization)
  neck circumference,
factors of internal vein jugular catheterization success | Baseline (Before catheterization)
  internal juguler vein depth
factors of internal vein jugular catheterization success | Baseline (Before catheterization)
  internal vein diameter
factors of internal vein jugular catheterization success | Baseline (Before catheterization)
  pleth variability index

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Zonguldak Bülent Ecevit University Faculty of Medicine, Kozlu, Esenköy
  - Zongulak Bülent Ecevit University, Zonguldak, Kozlu

IPD SHARING:
Plan to Share IPD: No